CLINICAL TRIAL: NCT02990533
Title: Translating Muscle Anabolic Strategies Into Interventions to Accelerate Recovery From Hospitalization in Geriatric Patients
Brief Title: Muscle Anabolic Interventions to Accelerate Recovery From Hospitalization in Geriatric Patients
Acronym: GRAMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-0146
Record Dates: First submitted 2016-10-25; First posted 2016-12-13 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Aging
MeSH Terms: interventions — Testosterone; testosterone enanthate; Whey Proteins; Sodium Chloride; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo Supplement Placebo Injection
  Interventions: Other: Placebo Injection; Other: Placebo supplement
- Testosterone (Experimental): Placebo Supplement Testosterone Injection
  Interventions: Drug: Testosterone; Other: Placebo supplement
- Protein Supplement (Experimental): Protein Supplement Placebo Injection
  Interventions: Dietary Supplement: Protein Supplement; Other: Placebo Injection
- Protein Supplement + Testosterone (Experimental): Protein Supplement Testosterone Injection
  Interventions: Drug: Testosterone; Dietary Supplement: Protein Supplement

INTERVENTIONS:
Drug: Testosterone
  Other Names: testosterone enanthate
  Arms: Protein Supplement + Testosterone; Testosterone
Dietary Supplement: Protein Supplement
  Other Names: whey protein
  Arms: Protein Supplement; Protein Supplement + Testosterone
Other: Placebo Injection
  Other Names: saline
  Arms: Placebo; Protein Supplement
Other: Placebo supplement
  Other Names: maltodextrin
  Arms: Placebo; Testosterone

SUMMARY:
The goal of this pilot study is to collect preliminary data on the feasibility and effect size of interventions to modify the physiological recovery trajectory from hospitalization in community dwelling older adults.

DETAILED DESCRIPTION:
The purpose of this pilot study is to test the feasibility and effect size of interventions to modify the physiological recovery trajectory from hospitalization in community dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the UTMB hospital
* Aged 65 years or older
* Self-reported ability (with or without the aid of an assistive device) to walk across a small room two weeks prior to hospitalization
* Alert and oriented x3 by a physician on H&P.
* Discharged "to home" at hospital discharge. Participation in the study will be terminated in those subjects not discharged to home after hospital stay.

Exclusion Criteria:

* A Nursing home resident or hospice care patient
* Uncontrolled blood pressure (systolic >170, or diastolic > 100)
* New onset motor disability that prevents walking at the time of baseline testing (stroke with motor disability, lower limb orthopedic dx)
* End stage renal disease
* AST/ALT 2.5 times above the normal limit
* Recent (within 3 months) or current treatment with anabolic steroids.
* History of breast or prostate cancer
* Palpable prostate nodule or induration or prostate specific antigen (PSA) ≥ 4 ng/ml (PSA ≥ 3 ng/ml in men at high risk of prostate cancer)
* Hematocrit ≥ 50%
* Any other condition or event considered exclusionary by the PI and faculty physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Physical Performance | Change from Baseline to 30-day Followup
  Short Physical Performance Battery (SPPB) scale, 0-12 points. 0=disabled; 12=high performance

SECONDARY OUTCOMES:
Handgrip Strength | Change from Baseline to 30-day Followup
  strength by handheld dynamometer, kg
Physical Activity Level | Change from Baseline to 30-day Followup
  Number of daily steps
30 day re-admission | 30 days post-discharge
  Readmission within 30 days of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Study Chair — UTMB
Locations (1):
- Jennie Sealy Hospital, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arentson-Lantz EJ, Boyle JT, Deer RR, Kokonda M, Bennetsen D, Carreon SA, Meers JM, Taffet G, Vahidy FS, Agarwal KS, Volpi E, Nowakowski S. Association of Sleep Disturbance and Physical Functioning Following Acute Hospitalisation in Older Adults. J Sleep Res. 2025 Nov 29:e70252. doi: 10.1111/jsr.70252. Online ahead of print. PMID 41316872